CLINICAL TRIAL: NCT03145051
Title: Prospective, Randomized, Cross-over, Multicenter, Trial Comparing the Efficacy and Tolerability of Nasal Irrigation With Respimer® Netiflow® Mineral Salts Solution Versus Saline Among Patients With Cystic Fibrosis and Suffering From Chronic Rhinosinusitis
Brief Title: Efficacy of Nasal Irrigation With Respimer® Netiflow® vs Saline Among Patients With Cystic Fibrosis and Chronic Rhinosinusitis
Acronym: Respire
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratoire de la Mer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Laboratoiredelamer
Record Dates: First submitted 2016-11-15; First posted 2017-05-09 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Chronic Rhinosinusitis; Cystic Fibrosis
Keywords: saline solution; minerals; cystic fibrosis; chronic rhinosinusitis; nasal irrigation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respimer Netiflow mineral salts solution (Experimental): Nasal irrigation with Respimer Netiflow mineral salts solution, 4 times/day during 8 weeks using Respimer Netiflow class I medical device
  Interventions: Other: Respimer Netiflow
- Saline solution (Active Comparator): Nasal irrigation with saline solution , 4 times/day during 8 weeks using Respimer Netiflow class I medical device
  Interventions: Other: Saline solution

INTERVENTIONS:
Other: Saline solution — a nasal irrigation care
  Other Names: nasal irrigation care
  Arms: Saline solution
Other: Respimer Netiflow — a nasal irrigation care
  Other Names: nasal irrigation care
  Arms: Respimer Netiflow mineral salts solution

SUMMARY:
Prospective, randomized, cross-over, multicenter, trial comparing the efficacy and tolerability of nasal irrigation with Respimer® mineral salts solution versus saline solution both administered with Respimer® Netiflow® medical device among patients aged ≥ 11 years and older with cystic fibrosis and suffering from chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

* • Patient with Cystic Fibrosis with or without lung transplant;

  * Patients with allergic chronic rhino sinusitis or no allergic diagnosed by the clinical investigator on the basis of the following signs in variable combination: nasal congestion, headache, sneezing, itchy nose and eyes, runny nose, nosebleeds and nasal crusts, redness and eye discharge present more than 3 months per year.
  * Patient treated on an outpatient basis;
  * Patient agreeing not to take sea baths for the duration of the study;
  * Patient agreeing to respect the procedures for conducting the study, in particular the washout period and follow-up visits;
  * Patient capable of understanding and self-completing the questionnaires;
  * For juvenile patients, the holder (s) of parental authority have accepted the participation of the young person (by signing the informed consent after having taken note of the information note)
  * Member or beneficiary of a social security program

Exclusion Criteria:

* Patients with significant obstruction of the nasal passages due to:
* a mucocele,
* polyposis causing nasal obstruction> 90% or
* severe malformation of the septum causing a nasal obstruction> 90% in whom surgical treatment is recommended;

  * Patients with signs of severity that may require hospitalization, such as: severe impairment of general health, dyspnoea with cyanosis, high fever (> 40 ° C).
  * Patients requiring corticosteroid therapy during the study, with the exception of patients who received pulmonary transplant and were treated with oral corticosteroids at no more than 0.2 mg / kg / day.
  * Patients with known systemic immunodeficiency status with the exception of patients receiving pulmonary transplantation and immunosuppressed.
  * Patient pregnant (urine test) or without effective contraception (birth control pill, contraceptive patch, contraceptive implant, vaginal ring, intrauterine device or intrauterine device, male condom).
  * Nursing patient.
  * Patient with a contraindication to nasal irrigations as defined in the product leaflet.

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life among subjects undergoing nasal irrigation with Respimer® Netiflow® mineral salts solution compared to saline solution between inclusion and the end of treatment period. | over an 8 weeks period
  Quality of life to be assessed over an 8 weeks period of nasal wash using SNOT-20 questionnaire

SECONDARY OUTCOMES:
Clinical status evolution among subjects undergoing nasal irrigation with Respimer® Netiflow® mineral salts solution to saline solution between inclusion and the end of treatment period. | over an 8 weeks period
  Clinical status to be assessed after 4 and 8 weeks of nasal wash using Lund-Kennedy Symptomatic Score (LKSS)
Endoscopic status evolution among subjects undergoing nasal irrigation with Respimer® Netiflow® mineral salts solution to saline solution between inclusion and the end of treatment period. | over an 8 weeks period
  Endoscopic status to be assessed after 4 and 8 weeks of nasal wash using Lund-Kennedy Endoscopic Score (LKES)
Mucociliary transport change among subjects undergoing nasal irrigation with Respimer® Netiflow® mineral salts solution to saline solution between inclusion and the end of treatment period. | over an 8 weeks period
  Mucociliary transport to be assessed after 4 and 8 weeks of nasal wash using saccharine test
Evolution of nasal bacterial pathogens among subjects undergoing nasal irrigation with Respimer® Netiflow® mineral salts solution to saline solution between inclusion and the end of treatment period. | over an 8 weeks period
  Evolution of nasal bacterial pathogens to be assessed by bacteriologic swab within ethmoid nasal cavities after 4 and 8 weeks of nasal wash
Patient treatment acceptance of nasal irrigation with Respimer® Netiflow® medical device | over an 8 weeks period
  Patient treatment acceptance to be assessed by Morisky score after 4 and 8 weeks of nasal wash
Occurrence of adverse events : taste impairment, epistaxis, nasal irritations, nasal burning | over an 8 weeks period
  Adverse events to be assessed based on vigilance tracking during the whole study period

CONTACTS AND LOCATIONS:
Locations (1):
- ORL et Chirurgie Cervico-faciale Centre Hospitalier Intercommunal (CHI) de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No